CLINICAL TRIAL: NCT06073262
Title: Investigation of the Effect of Low Back Pain Level on Symptoms in Individuals With Chronic Consipation
Brief Title: Investigation of Low Back Pain Level on Symptoms in Chronic Consipation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-5856
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain; Constipation
Keywords: pain; Low Back Pain; Constipation
MeSH Terms: conditions — Low Back Pain; Constipation; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-specific low back pain individual with chronic consipation
- Individual without low back pain with chronic consipation

SUMMARY:
Consipation is the most common digestive complaint in the general population

DETAILED DESCRIPTION:
Chronic constipation and low back pain are two common and often co-existing health conditions that affect millions of people worldwide. On the surface, these conditions appear to be unrelated and are associated with different anatomical sites (gastrointestinal tract and musculoskeletal system). However, a growing body of research is beginning to shed light on the complex interplay between chronic constipation and low back pain, highlighting potential links between these seemingly disparate health conditions. Common etiologic factors such as neuromuscular function, chronic inflammation and lifestyle-related variables are known to exist

ELIGIBILITY:
Inclusion Criteria:

* 18-65 ages
* Rome III diagnostic criteria

Exclusion Criteria:

* Severe heart or kidney diseaseprevious gastrointestinal, spinal or pelvic surgery other than cholecystectomy, hysterectomy or appendectomy neurological diseases such as
* Multiple sclerosis, stroke, Parkinson's disease or spinal injury,
* Impaired awareness (mini-mental score < 15),
* Legal blindness, pregnancy,
* Rectal prolapse
* Anal fissure and altered constipation and diarrhea pattern.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study, Rome III diagnostic criteria, which is the most commonly used diagnostic method, will be used to determine constipation status. According to the Rome III diagnostic criteria, the following symptoms must have been present for the last 3 months and these symptoms must have started at least 6 months before the diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Bristol Stool Scale | one day
  Lewis and Heaton classified the type of stool in 7 different groups in the scale. In the Bristol Stool Scale, the transit time of stool through the intestine is evaluated over seven different stool types. According to BGS, 1-2 points are shown as "hard stool", 3-4-5 points as "normal stool" and 6-7 points as "soft-watery stool (diarrhea)".
Pelvic Pain Impact Questionnaire | one day
  The questionnaire for clinical assessment of the impact of pelvic pain on women consists of 10 questions. However, the first 8 questions are scored. The range of scores to be obtained from the questionnaire varies between 1- 32. As the score value to be obtained from the questionnaire increases, the degree of functional limitation of pelvic pain on the person increases.
Constipation Severity Scale | one day
  Constipation Severity Scale (CSS) is a scale for determining the frequency, intensity and difficulty/difficulty during defecation. The scale includes 16 questions.
  The score that can be obtained from the DT sub-dimension is between 0-28, the score that can be obtained from the CBT sub-dimension is between 0-29, and the score that can be obtained from the Pain sub-dimension is between 0-16. The minimum total score that can be obtained from the KCS is 0 and the maximum score is 73. A high score on the scale indicates that the symptoms are serious. The highest score that can be obtained from the five-point Likert-type scale is 140 and the lowest score is 28. It is thought that quality of life is negatively affected as the scores obtained from the scale increase
Disability level | one day
  The Oswestry Disability Index is a commonly used outcome measure to detect perceived disability in patients with low back pain (12). This index consists of 10 items, 8 related to activities of daily living and 2 related to pain. Each item is scored from 0-5 and the total score is expressed as a percentage, with higher scores corresponding to more disability). Increasing scores on the Oswestry Disability Index indicate a higher level of disability.
Autonomic nervous system device (Polar H10) | one day
  The Polar H10 device is a heart rate sensor with the gold standard in high precision and accuracy that comes with a wearable chest strap. It can connect to multiple training devices via Bluetooth and ANT+. The device comes with a soft, adjustable sensor that contacts the chest to capture heart rate in real time.
  The study will evaluate the autonomic nervous system with the Polar H10 device. The data will be recorded by connecting the device to a smart phone via bluetooth and the software supported by the device will be used to analyze the data. The participant will be in a sitting position and a measurement will be made for 1 minute. In order for the device to make an accurate measurement, the electrode surface must be wetted before each measurement. The subject should not talk or move during the measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)